CLINICAL TRIAL: NCT03185897
Title: A Global Epidemiologic Study to Determine the Prevalence of Neutralizing Antibodies and Related Adaptive Immune Responses to Adeno-Associated Virus (AAV) in Adults With Hemophilia
Brief Title: Global Epidemiologic Study of Preexisting Immunity to AAV in Adults With Severe Hemophilia
Status: Completed | Type: Observational
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: 201601
Record Dates: First submitted 2017-05-31; First posted 2017-06-14 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Hemophilia A; Hemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — Seroepidemiologic Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemophilia A: Participants with hemophilia A
  Interventions: Other: Non-treatment, seroprevalence
- Hemophilia B: Participants with hemophilia B
  Interventions: Other: Non-treatment, seroprevalence

INTERVENTIONS:
Other: Non-treatment, seroprevalence — Non-treatment study examining the prevalence of preexisting immunity to adeno-associated virus (AAV)

SUMMARY:
Assess the seroprevalence of neutralizing antibodies (NAb) to AAV in adults with severe hemophilia A (coagulation factor VIII [FVIII] <1%) or moderately severe to severe hemophilia B (coagulation factor IX [FIX] ≤2%).

ELIGIBILITY:
Inclusion Criteria:

1. Participant is male between 18 and 75 years old at the time of screening.
2. Established severe hemophilia A (plasma Factor VIII (FVIII) activity <1%) or B (plasma Factor IX (FIX) activity ≤2%).
3. Provision of signed informed consent form (ICF).
4. Participant is willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

1. Bleeding disorder(s) other than hemophilia A or B.
2. Personal laboratory evidence of having developed inhibitors to FVIII or FIX protein at any time (≥0.6 Bethesda Units [BU] on any single test).
3. Currently receiving systemic immunosuppressive therapy, cytotoxic chemotherapy, immunoglobulin therapy, or monoclonal antibody therapy.
4. Received systemic antiviral and/or interferon therapy within 30 days of blood draw, with the exception of treatment for human immunodeficiency virus (HIV).
5. Currently receiving ribavirin and/or interferon based therapy for active hepatitis C virus (HCV).
6. Received immunoglobulin therapy or plasma infusion within 120 days of the blood draw.
7. Has a known immune deficiency other than HIV.
8. Has lymphocyte or plasma cell malignancies.
9. Participant is a family member or employee of the investigator.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemophilia A and hemophilia B patients who receive treatment at Hemophilia Treatment Centers.
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
Prevalence of neutralizing antibodies (NAb) - Baseline visit | Baseline visit
  Prevalence of NAb to naturally occurring adeno-associated virus (AAV) serotypes
Prevalence of neutralizing antibodies (NAb) - Year 1 Visit | Year 1 visit
  Prevalence of NAb to naturally occurring adeno-associated virus (AAV) serotypes
Prevalence of neutralizing antibodies (NAb) - Year 2 Visit | Year 2 visit
  Prevalence of NAb to naturally occurring adeno-associated virus (AAV) serotypes
Prevalence of neutralizing antibodies (NAb) - Year 3 Visit | Year 3 visit
  Prevalence of NAb to naturally occurring adeno-associated virus (AAV) serotypes

SECONDARY OUTCOMES:
Prevalence of NAb to AAV including AAV2 and AAV8 | Baseline visit, Year 1 visit, Year 2 visit, and Year 3 visit
  Prevalence of neutralizing antibodies (NAb) to adeno-associated virus (AAV) including AAV2 and AAV8
Prevalence of binding antibodies to AAV, including AAV8 and AAV2 | Baseline visit, Year 1 visit, Year 2 visit, and Year 3 visit
  Prevalence of binding antibodies to adeno-associated virus (AAV), including AAV8 and AAV2
T-cell mediated immune response to AAV8 | Baseline visit, Year 1 visit, Year 2 visit, and Year 3 visit
  T-cell mediated immune response to AAV8

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (23):
- United States (7):
  - Orthopaedic Hemophilia Treatment Center, Los Angeles, California
  - University of Colorado Hemophilia & Thrombosis Center, Aurora, Colorado
  - Michigan State University, East Lansing, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Gulf States Hemophilia and Thrombophilia Center, Houston, Texas
  - University of Washington, Seattle, Washington
- AKH - Medizinische Universität Wien, Vienna, Austria
- France (6):
  - Hôpital Morvan, Brest
  - Groupement Hospitalier Est- Hôpital Louis Pradel, Bron
  - Groupement Hospitalier Sud - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hopital Jeanne de Flandre - CHU Lille, Lille
  - Hôpital de la Timone, Marseille
  - CHU de Nantes Site Hotel Dieu, Nantes
- Germany (2):
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt
- Italy (4):
  - Presidio Ospedaliero di Castelfranco Veneto, Castelfranco Veneto
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale San Bortolo di Vicenza, Vicenza
- Spain (3):
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fc54db2bf003ab45d07